CLINICAL TRIAL: NCT06521255
Title: A Randomized, Multi-center, Phase 3 Study of Tafasitamab and Lenalidomide in Combination With Gemcitabine and Oxaliplatin Versus Rituximab in Combination With Gemcitabine and Oxaliplatin in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: Evaluate the Safety and Efficacy of Tafasitamab and Lenalidomide in Combination With Gemcitabine and Oxaliplatin Versus Rituximab in Combination With Gemcitabine and Oxaliplatin in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00903
Record Dates: First submitted 2024-07-15; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-06

CONDITIONS: DLBCL
MeSH Terms: interventions — tafasitamab; Lenalidomide; Gemcitabine; Oxaliplatin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tafasitamab and lenalidomide in combination with gemcitabine and oxaliplatin (Experimental)
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide; Drug: Gemcitabine; Drug: Oxaliplatin
- Rituximab in combination with gemcitabine and oxaliplatin (Active Comparator)
  Interventions: Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Rituximab

INTERVENTIONS:
Drug: Tafasitamab — Tafasitmab was infused intravenously
  Arms: Tafasitamab and lenalidomide in combination with gemcitabine and oxaliplatin
Drug: Lenalidomide — Lenalidomide orally
  Arms: Tafasitamab and lenalidomide in combination with gemcitabine and oxaliplatin
Drug: Gemcitabine — Gemcitabine was infused intravenously
Drug: Oxaliplatin — Oxaliplatin was infused intravenously
Drug: Rituximab — Rituximab was infused intravenously.
  Arms: Rituximab in combination with gemcitabine and oxaliplatin

SUMMARY:
This is a Randomized, Multi-center, Phase 3 Study of Tafasitamab and Lenalidomide in Combination with Gemcitabine and Oxaliplatin versus Rituximab in Combination with Gemcitabine and Oxaliplatin in Patients with Relapsed/Refractory Diffuse Large B-Cell Lymphom

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years and older.
2. One of the histologies of DLBCL confirmed by participated sites below with，not otherwise specified;T-cell/histiocyte-rich large B-cell lymphoma;Epstein-Barr virus (EBV) positive DLBCL (EBV-positive DLBCL); Composite lymphoma with a DLBCL component with a subsequent DLBCL relapse; Disease transformed from an earlier diagnosis of low-grade lymphoma into DLBCL with DLBCL treatment failure.
3. Availability of tumor tissue biopsied post last line of therapy and prior to current study treatment for the patients enrolled in safety and tolerability stage.
4. Relapsed/refractory (R/R) DLBCL, at least one (≥1) but no more than three (≤3) line of prior systemic therapies.
5. Patients who have not received high dose therapy/stem cell transplantation (HDT/SCT) must be ineligible for HDT/SCT.
6. At least one measurable site of disease per CT or magnetic resonance imaging (the longest axis of the lymph node lesion is > 1.5 cm, and the longest diameter of the extra-nodal lesion is > 1.0 cm).
7. ECOG PS score of 0 to 2.
8. Subject must have adequate organ functions, and the laboratory values comply with the protocol requirements.
9. Life expectancy of ≥ 3 months.
10. Informed consent before screening and can understand and comply with the requirements of the study.

Exclusion Criteria:

1. Existing or prior history of other malignant tumor within 3 years, except for those who have received curative treatment.
2. Current or history of central nervous system (CNS) lymphoma.
3. Known high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements.
4. Primary mediastinal B-cell lymphoma.
5. History of allogeneic stem-cell transplantation.
6. Prior exposure to anti-CD19 treatment, and (or) failed with gemcitabine plus platinum-based agent combination therapy.
7. Current toxicity of ≥ Grade 2 from prior anti-cancer therapy (except for alopecia, neutrophil, hemoglobin and platelets).
8. Clinically significant cardiovascular disease or nervous system disease.
9. History of deep venous thrombosis/embolism, threatening thromboembolism or known thrombophilia or are at a high risk for a thromboembolic event in the opinion of the investigator and who are not willing/able to take venous thromboembolic event prophylaxis during the entire treatment period.
10. Uncontrolled systemic infection requiring parenteral intravenous anti-infective therapy.
11. Known human immunodeficiency virus (HIV), or serologic status reflecting active hepatitis B or C infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity（DLT）and other adverse events (AEs) of tafasitamab and lenalidomide in combination with GemOx (TL-GemOx) assessed using CTCAE v5.0 | within 28 days after therapy initiation
PFS assessed by IRC according to Lugano 2014 | 1-3 years approximately

SECONDARY OUTCOMES:
Objective Response Rate (ORR) according to investigator. | 1-3 years approximately
Complete Response Rate (CRR) according to investigator. | 1-3 years approximately
Duration of Response (DOR) according to investigator. | 1-3 years approximately
Progression free survival (PFS) assessed by investigator according to the Lugano 2014 | 1-3 years approximately
Time to response (TTR) | 1-3 years approximately
Overall Survival (OS) | 1-3 years approximately
Time to next treatment (TTNT) | 1-3 years approximately
Adverse events assessed by CTCAE version 5.0 criteria. | 1-3 years approximately
Quality of life assessment: Patient-reported outcomes (PROs) on happiness and general health status based on Functional Assessment of Cancer Therapy-Lymphoma (FACT-Lym) | 1-3 years approximately
Quality of life assessment: Patient-reported outcomes (PROs) on happiness and general health status based on EuroQol five dimensions questionnaire (EQ-5D-5L) | 1-3 years approximately

CONTACTS AND LOCATIONS:
Locations (20):
- China (20):
  - Beijing Hospital, Beijing
  - The First Hospital Of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - Chenzhou No.1 People's Hospital, Chaozhou
  - Sichuan Province People's Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Guangdong General Hospital, Guangzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Hangzhou First People's Hospital, Hangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Shandong Cancer Hospital and Institute, Jinan
  - Jiangxi Cancer Hospital, Nanchang
  - The First Affiliated Hospital of Nanchang University, Nanjing
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Tianjin First Central Hospital, Tianjin
  - Xinjiang Medical University Affiliated Cancer Hospital, Ürümqi
  - The First Affiliated Hospital Wenzhou Medical University, Wenzhou
  - Union Hospital Tongji Medical College, Wuhan
  - Henan Cancer Hospital, Zhengzhou